CLINICAL TRIAL: NCT06839677
Title: PERCEPTION of QUALITY of LIFE in PATIENTS UNDERGOING ENDOSCOPIC VERTICAL GASTROPLASTY: a DESCRIPTIVE EXPLORATORY STUDY
Acronym: SATIBAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Massari Chiara, Research nurse, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7204
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Endoscopy; Quality of Life of Patients; ENDOSCOPIC VERTICAL GASTROPLASTY; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Prospective multi-centre exploratory descriptive observational study, survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: semi-structured interview on Microsoft Teams — Data will be collected through a single semi-structured interview on Microsoft Teams, audio recorded and transcribed in full, and analysed using NVivo V1.6.2.32. Participants' statements will be categorised into semantic categories and subsequently refined into sub-themes and themes through an iterative process.

SUMMARY:
An emerging alternative to bariatric surgery for the treatment of obesity is bariatric endoscopic gastroplasty (gve), which offers a less invasive approach with fewer complications. however, the weight loss achieved through this technique is generally lower than that achieved with traditional bariatric surgery, leaving the impact on patients' quality of life uncertain. the aim of this multicentre exploratory descriptive study is to investigate the perception of the quality of life of patients with obesity undergoing gve, conducted at the complex operative unit of surgical digestive endoscopy of the university policlinico Agostino Gemelli IRCCS foundation as the promoting centre. italian patients over 18 years old, in post-gve follow-up for at least six months, with access to and familiarity with a computer or tablet will be included. data will be collected via a single semi-structured interview on microsoft teams, audio recorded and transcribed in full, and analysed using nvivo v1.6.2.32. participants' statements will be categorised into semantic categories and subsequently refined into sub-themes and themes through an iterative process.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients older than 18 years.
* Treatment: Patients who have undergone GVE surgery and have been in post- surgery for at least six months.
* Access and technological competence: Patients who have a computer or tablet at home and are familiar with their use.
* Informed consent: Patients who are able to understand and give informed consent informed consent to participate in the study.
* Language comprehension: Patients who have a good understanding of the language Italian language, both written and spoken, to ensure correct completion and understanding of the informed consent and the study instructions.

Exclusion Criteria:

* Patients who have been enrolled in experimental studies involving additional procedures during GVE will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The perception of quality of life will be investigated through specific questions | From treatment with GVE to ineterview. At least six months
  The perception of quality of life will be investigated through specific questions regarding: general well-being and satisfaction with different aspects of daily life, including personal satisfaction and perception of one's own body after the procedure, allowing participants to freely express their perceptions, concerns and wishes regarding their post-operative experience after GVE.
  Overall satisfaction with the GVE procedure.

SECONDARY OUTCOMES:
Analysis of positive and negative experiences post-GVE | From treatment with GVE to ineterview. At least six months
  Analysis of positive and negative experiences with post-GVE to identify areas for improvement in the management of the patient undergoing GVE.